CLINICAL TRIAL: NCT02412631
Title: Varenicline and Lorcaserin for Smoking Cessation and Weight Gain Prevention
Brief Title: Addressing Post Cessation Weight Gain
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lorcaserin removed from market
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., Associate Professor, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-005230; 1K23DA037299-01A1 (NIH); 14-005682 (Other: Mayo Clinic)
Record Dates: First submitted 2015-03-12; First posted 2015-04-09 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Obesity; Smoking Cessation
MeSH Terms: conditions — Obesity; Smoking Cessation | interventions — lorcaserin; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline plus placebo (Placebo Comparator): Subjects will receive open label varenicline (12 weeks) plus a placebo for lorcaserin (24 weeks)
  Interventions: Drug: Varenicline; Drug: Placebo
- Varenicline plus lorcaserin (Experimental): Subjects will receive open label varenicline (12 weeks) plus lorcaserin (24 weeks)
  Interventions: Drug: lorcaserin; Drug: Varenicline

INTERVENTIONS:
Drug: lorcaserin — lorcaserin is an FDA-approved weight loss medication for overweight and obese patients
  Other Names: Belviq
  Arms: Varenicline plus lorcaserin
Drug: Varenicline — Chantix is an FDA approved medication for smoking cessation
  Other Names: Chantix
Drug: Placebo — Placebo for lorcaserin
  Arms: Varenicline plus placebo

SUMMARY:
Some individuals smoke with the perception that smoking helps control body weight. Smokers gain an average of as much as 10 pounds in the months following smoking abstinence, with heavier and more-dependent smokers gaining more weight. T The Mayo Clinic Nicotine Research Program will randomize 100 nondiabetic, overweight or obese adult smokers to active lorcaserin or placebo for 24 weeks; all of the subjects will receive open-label varenicline for 12 weeks. The purpose of this study is to assess the efficacy of a 24-week course of lorcaserin for decreasing weight gain after stopping smoking.

DETAILED DESCRIPTION:
This will be a randomized, placebo-controlled, parallel-group clinical trial. Nondiabetic, overweight and obese adult smokers will be randomized to one of three arms:

* lorcaserin for 24 weeks in combination with varenicline for 12 weeks;
* placebo for 24 weeks in combination with varenicline for 12 weeks;

We will assess the following:

* changes in weight and Weight Concern
* 7-day point-prevalence smoking abstinence weekly through week 24 and prolonged smoking abstinence at 24 and 52 weeks. Subjects will have a target quit date 8 days after starting medication.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered for inclusion if they meet all of the following

1. ≥18 years and ≤65 years of age;
2. smoked ≥10 cigarettes/day for the past 6 months;
3. Body Mass Index of 27-39.9 kg/m2;
4. motivated to stop smoking;
5. weight concerned as shown with the Weight Concern Scale;
6. able to participate fully in all aspects of the study;
7. understand and signed the study informed consent.
8. Subject is in good health as determined by the clinical investigators.

Exclusion Criteria:

Subjects will be ineligible for participation if they have any of the following:

1. current nonspecific suicidal thoughts or a lifetime history of a suicidal attempt (defined by the Columbia-Suicide Severity Rating Scale as a "potentially self-injurious act committed with at least some wish to die, as a result of act.");
2. current moderate or severe depression as assessed by a score of ≥16 on the Center for Epidemiology Studies-Depression;
3. a lifetime history of psychosis, bipolar disorder or schizophrenia;
4. use of anti-psychotic medication within the past 30 days;
5. use of weight-loss medications within the past 30 days or current participation in a program specifically designed to help with weight loss;
6. weight fluctuations of 20 pounds or more in the past 6 months (self-report);
7. use of any treatments for tobacco dependence within the past 30 days;
8. use of an investigational drug within the past 30 days;
9. recent history (past 3 months) of abuse of or dependence on a substance other than tobacco. Including: heavy alcohol consumption (If male, drinking > 4 alcoholic beverages per day for past month and if female, drinking > 3 alcoholic beverages per day for past month); use of cocaine, heroin, club drugs (i.e., methylenedioxymethamphetamine(MDMA)/"ecstasy"), methamphetamine, or hallucinogens (e.g., LSD) at any time during the past 3 months; and use of marijuana on a weekly basis for the past 3 months
10. current use of triptans, monoamine oxidase inhibitors, selective serotonin reuptake inhibitors (SSRI), selective serotonin-norepinephrine re-uptake inhibitors (SNRI), dextromethorphan, tricyclic antidepressants (TCA), bupropion, lithium, tramadol, tryptophan, and St. John's Wort, or any other medication known to involve the serotonergic neurotransmitter system (see human subjects section);
11. uncontrolled hypertension (systolic >160 mm Hg and/or diastolic >100 mm Hg) documented on 2 separate occasions;
12. current use of medications known to interact with varenicline or lorcaserin. These can include benzodiazepines, narcotics, anti-epileptics;
13. another household member or relative participating in the study;
14. known diabetes;
15. a known allergy to varenicline or lorcaserin.
16. Women who are pregnant or lactating, or who are of childbearing potential and are likely to become pregnant during the medication phase but are not willing to use a reliable form of contraception, will also be excluded. Reliable forms of contraception include oral contraception, diaphragm or condom (with spermicide), injections, intrauterine device, surgical sterilization, and abstinence.
17. Has an unstable medical condition as determined by the physician investigator
18. Subject describes having a medical history of: a) unstable angina; b) myocardial infarction within the past 3 months; c) coronary angioplasty or d) an untreated cardiac dysrhythmia.
19. Subject currently has cancer [excluding non-melanoma skin cancer] not in remission
20. Known history of seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T Hurt, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurt RT, Croghan IT, Schroeder DR, Choi DS, Fischer K, Fokken S, Ebbert JO. Varenicline and Lorcaserin for Smoking Cessation and Weight Gain Prevention: A Randomized Clinical Trial. Mayo Clin Proc Innov Qual Outcomes. 2022 Sep 21;6(5):465-474. doi: 10.1016/j.mayocpiqo.2022.01.004. eCollection 2022 Oct. PMID 36160639
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between June 16th, 2016 to January 22nd, 2020. Recruitment was in three phases: initial phone pre-screen, followed by a consent visit and study screen, and finally a randomization visit. All visits took place at a medical clinic.
Period: Overall Study
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin
Started | 44 | 40
Completed | 18 | 16
Not Completed | 26 | 24
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 5 | 9
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Early stop by FDA | 5 | 2
Not completed — Unspecified reason | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin | Total
Number analyzed (Participants) | 44 | 40 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (9.05) | 43.4 (10.98) | 42.3 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 42 | 40 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 37 | 78
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Baseline Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 17.2 (5.59) | 17.9 (5.96) | 17.5 (5.75)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 91.8 (15.46) | 93.4 (14.7) | 92.6 (15.03)

OUTCOME MEASURES:

1. Primary Outcome: Post Cessation Weight Gain (kg)
Description: weight (kg) change from baseline to week 24 among subjects who meet criteria for prolonged smoking abstinence at week 24
Time Frame: 24 weeks
Population: Restricted to those who met criteria for prolonged abstinence at week 24.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin
Number analyzed (Participants) | 13 | 8
kg | 0.7 (8.38) | 2.2 (2.07)

2. Secondary Outcome: BMI
Description: BMI change from baseline to week 24
Time Frame: 24 weeks
Population: Restricted to those who met criteria for prolonged abstinence at week 24.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin
Number analyzed (Participants) | 13 | 8
kg/m^2 | 0.5 (2.91) | 0.8 (0.72)

3. Secondary Outcome: Smoking Abstinence
Description: Lorcaserin combined with open label varenicline will be evaluated for improved smoking abstinence compared to placebo
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin
Number analyzed (Participants) | 44 | 40
Participants | 13 | 8

4. Secondary Outcome: Waist Circumference
Description: Waist Circumference change from baseline to week 24
Time Frame: 24 weeks
Population: Restricted to those who met criteria for prolonged abstinence at week 24.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin
Number analyzed (Participants) | 13 | 8
cm | 0.8 (7.60) | -0.1 (2.97)

5. Secondary Outcome: Fat Mass
Description: Body Fat difference from baseline to week 24.
Time Frame: 24 weeks
Population: Restricted to those who met criteria for prolonged abstinence at week 24.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin
Number analyzed (Participants) | 13 | 8
kg | 0.4 (7.12) | 2.2 (2.74)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected throughout the 24 week study period.
Description: Reported AEs were included in this section.
Arm/Group | Varenicline Plus Placebo | Varenicline Plus Lorcaserin
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/40
Other Adverse Events (participants affected / at risk) | 21/44 | 18/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline Plus Placebo (N=44) | Varenicline Plus Lorcaserin (N=40)
Headache (Nervous system disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 2 | 5
GI (Gastrointestinal disorders) | 5 | 4 — Includes upset stomach, abdominal pain, bloating, and diarrhea.
Nausea (Gastrointestinal disorders) | 8 | 5
Sleep disorders (General disorders) | 9 | 7 — Includes sleep disorders and vivid dreams
Mood (Nervous system disorders) | 0 | 3 — Includes irritability and depression
Dry Mouth (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT02412631/Prot_SAP_000.pdf